CLINICAL TRIAL: NCT03582189
Title: A Feasibility Study of Magnetic Resonance Imaging (MRI) as a Platform for Image Guidance and Adaptive Radiation Therapy in Patients With Liver or Pancreatic Cancer
Brief Title: MR Guidance for Liver and Pancreas
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 18-5176
Record Dates: First submitted 2018-05-01; First posted 2018-07-10 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Magnetic Resonance Imaging
Keywords: Liver Cancer; Pancreatic Cancer; Radiation
MeSH Terms: conditions — Liver Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pancreatic Cancer: Approximately 10 patients with pancreatic cancer will be enrolled to the study with the primary aim of determining the feasibility of using off-line MRI-guidance during the course of radiation treatment
  Interventions: Other: MRI
- Liver Metastases: Approximately 10 patients with liver mets will be enrolled to the study with the primary aim of determining the feasibility of using off-line MRI-guidance during the course of radiation treatment
  Interventions: Other: MRI
- Hepatocellular carcinoma: Approximately 10 patients with HCC will be enrolled to the study with the primary aim of determining the feasibility of using off-line MRI-guidance during the course of radiation treatment
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — Patients who consent to this study will have an abdominal MRI prior to or immediately after each fraction of radiation treatment in the case of those patients that are undergoing SBRT or those receiving palliative treatment. On patients receiving definitive chemoradiation, an abdominal MRI will be performed prior to or immediately after radiation treatment once per week during the any five weeks of treatment

SUMMARY:
This is a single centre, single arm, prospective feasibility study that aims to see whether magnetic resonance imaging (MRI) as a source of image guidance before each radiation treatment fraction is feasible, and also if it may provide information that could potentially be used during the treatment to improve the radiation treatment plan.

Patients will have 5 MRIs with each of their RT sessions. If patients' RT treatment will consist of more than 5 fractions, only 5 MRIs will be done with any 5 RT fractions. Patients will be completing a short questionnaire at the end of each MRI. A patient questionnaire will also be completed at the end of the study to assess for patient satisfaction.

There will be 30 evaluable patients enrolled to the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older
* Diagnosed with locally advanced pancreatic cancer or hepatocellular carcinoma being considered for treatment with chemoradiation, long course RT, or SBRT with curative intent or palliative intent, planned for 5 or more RT fractions

Exclusion Criteria:

- Contraindications for MRI: ferromagnetic prosthesis, pacemaker / implanted defibrillator, claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with locally advanced pancreatic cancer or hepatocellular carcinoma being considered for treatment with chemoradiation, long course RT, or SBRT with curative intent or palliative intent, planned for 5 or more RT fractions
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-07-11 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction Survey | At study completion (day5 or week 5, depending on type of treatment)
  To evaluate patient satisfaction with the MR guidance process, a modified version of a questionnaire previously used at our institution will be performed at the end of the study
MRI-Anxiety Questionnaire | Prior to or before MR session 1 (day 1 or week 1, depending on type of treatment)
  This instrument will be used to evaluate patient related anxiety after each MR
MRI-Anxiety Questionnaire | Prior to or before MR session 2 (day 2 or week 2, depending on type of treatment)
  This instrument will be used to evaluate patient related anxiety after each MR
MRI-Anxiety Questionnaire | Prior to or before MR session 3 (day 3 or week 3, depending on type of treatment)
  This instrument will be used to evaluate patient related anxiety after each MR
MRI-Anxiety Questionnaire | Prior to or before MR session 4 (day 4 or week 4, depending on type of treatment)
  This instrument will be used to evaluate patient related anxiety after each MR
MRI-Anxiety Questionnaire | Prior to or before MR session 5 (day 5 or week 5, depending on type of treatment)
  his instrument will be used to evaluate patient related anxiety after each MR

CONTACTS AND LOCATIONS:
Overall Officials: Laura Dawson, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network - Princess Margaret Cancer Centre, Toronto, Ontario, Canada